CLINICAL TRIAL: NCT03913182
Title: Prospective,Single-arm,and Exploratory Phase II Clinical Study for the Efficacy of Apatinib in the Treatment of Recurrence or Metastasis of Esophageal Squamous Cell Carcinoma After Radical Resection
Brief Title: Apatinib in the Treatment of Recurrence or Metastasis of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Director, Head of esophageal surgery, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH0403
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Squamous Cell Carcinoma; Apatinib; Recurrence; Metastasis
Keywords: Esophageal squamous cell carcinoma; apatinib; recurrence; metastasis
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Recurrence; Neoplasm Metastasis | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: no special
Masking Description: no special
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib group (Experimental): apatinib：500mg po Qd
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — 500mg po Qd

SUMMARY:
It was difficult to obtain clinical benefits through traditional chemotherapy and radiotherapy for the patients who have recurrence or metastasis tumor even though they have received first-line chemotherapy or combined radiotherapy before, but failed.The aim of this study was to evaluate the safety and efficacy of apatinib, an anti-angiogenesis drug, in the treatment of patients with advanced esophageal squamous cell carcinoma who had recurrence or metastasis after radical resection

DETAILED DESCRIPTION:
Esophageal cancer is a common malignant tumor in China and its prognosis is poor. Its main treatment methods include surgery, radiotherapy and chemotherapy. However, the 5-year survival rate of esophageal cancer after operation is only about 40%. The main cause of treatment failure is postoperative recurrence and metastasis.The 2-year recurrence rate of esophageal cancer after radical operation was 50%, the median recurrence time was about 10 months and the 2-year survival rate was less than 15% for these patients.For patients with local recurrence, endoscopic submucosal resection, salvage resection and radiotherapy could be chosen. Palliative chemotherapy is another important method for patients with recurrence or metastasis who are not suitable for surgery or radiotherapy.Cisplatin combined with fluorouracil is a usually used first-line chemotherapy regimen, but the response rate is less than 30% and the median survival time is only about 6~10 months.There is no standard second-line treatment for patients who have failed first-line treatment. Over the past decade, the second-line treatment for esophageal cancer is mostly phase I and II studies. The reported objective remission rate(ORR) ranges from 2.8% to 45%, the median progression-free survival (PFS) ranges from 1.2 to 5.2 months and the median overall survival (OS) ranges from 3.7 to 11.4 months.Although some studies have shown that taxus-based second-line chemotherapy can bring a certain degree of remission to patients, irinotecan, gemcitabine and oxaliplatin can also be used as the second-line chemotherapy options for these patients, but the overall efficiency is low and disease progression occurs quickly.The median survival time of esophageal stent, nasal feeding nutrition support and gastrostomy is only 6 months, and the 1-year survival rate is generally less than 5%.The previous treatment options are few and the therapeutic effect is poor for the patients with locally advanced esophageal cancer who have received neoadjuvant chemotherapy combined with or without radiotherapy and adjuvant chemotherapy combined with or without radiotherapy after radical resection and those patients with persistent or new occurred recurrence and metastasis. At present, there is no consensus on the second-line treatment strategy for recurrent and metastasis esophageal squamous cell carcinoma after radical resection and there are various clinical options.Therefore, it is of great clinical significance to explore the second-line treatment strategy for these patients.

In recent years, with the development of molecular targeted therapy, it has been applied to the treatment of esophageal cancer, which is not only expected to ensure clinical efficacy, but also to reduce the adverse effects of amount of traditional chemotherapy and radiotherapy.At present, research on targeted therapy for esophageal cancer is gradually increasing. Targeted therapeutic drugs mainly include epidermal growth factor receptor(EGFR) inhibitors,vascular endothelial growth factor(VEGF) inhibitors, monoclonal antibodies, cyclooxygenase(COX) inhibitors and so on.Studies have confirmed that VEGF is highly expressed in the development of various malignant tumors including esophageal cancer, which may be closely related to tumor invasion and metastasis.As a VEGFR tyrosine kinase inhibitor, apatinib mainly treats malignant tumors by inhibiting VEGFR to exert anti-angiogenic effects.Previous studies have confirmed that apatinib was safe and effective in the treatment of advanced gastric cancer and adenocarcinoma of the gastroesophageal junction which was approved by China food and drug administration(CFDA).

In summary, it was difficult to obtain clinical benefits through traditional chemotherapy and radiotherapy for the patients who have recurrence or metastasis tumor even though they have received first-line chemotherapy or combined radiotherapy before, but failed.The aim of this study was to evaluate the safety and efficacy of apatinib, an anti-angiogenesis drug, in the treatment of patients with advanced esophageal squamous cell carcinoma who had recurrence or metastasis after radical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18;
2. ECOG score 0-2;
3. Postoperative pathology confirmed esophageal squamous cell carcinoma;
4. Have never received targeted therapy before;
5. Patients who had failed chemotherapy with platinum or paclitaxel regimens at least once in the past; Note: (1) At least one cycle of drug use, regardless of single or multiple drug combinations;(2) Neoadjuvant concurrent chemoradiotherapy, neoadjuvant chemotherapy or adjuvant chemotherapy are allowed;
6. According to RECIST version 1.1, there is at least one measurable lesion;
7. The estimated survival time is more than 3 months;
8. The main organs are functioning well, and the examination indicators meet the following requirements:

(1) Blood examination: Hemoglobin (>90 g/L) (no blood transfusion within 14 days);The neutrophil count (>1.5×109/L);Platelet count (> 80×109/L); (2)Biochemical examination:Total bilirubin<1.5×upper limit of normal (ULN);alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) are less than 2.5×ULN, ALT or AST are less than 5×ULN if liver metastasis occurred, and creatinine clearance is more than 50 ml/min (Cockcroft-Gault formula); 9.Sign the informed consent; 10.Good compliance, family members agreed to cooperate with survival follow-up;

Exclusion criteria

Subjects may not enter the trial with one of the following:

1. There were other malignant tumors at the same time, except cured skin basal cell carcinoma and cervical carcinoma in situ of cervix;
2. Pregnant or lactating women;
3. Participated in clinical trials of other drugs within one month;
4. Must be able to swallow tablets;
5. Any bleeding events with a severe grade of 3 or more in CTCAE 4.0 occurred within 4 weeks before screening;
6. Patients with central nervous system metastasis or a history of central nervous system metastasis before screening;
7. Patients with hypertension who can not be well controlled by a single anti-hypertensive drug (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg); those with a history of unstable angina pectoris; those newly diagnosed as angina pectoris within the first three months of screening or those with myocardial infarction within the first six months of screening; arrhythmia require long-term use of anti-arrhythmic drugs and cardiac insufficiency > Grade II (New York Heart Disease Association Grade) ;
8. Long-term nonunion of wounds or incomplete healing of fractures;
9. History of organ transplantation in the past;
10. Images show that the tumors have invaded important blood vessels or tumor was highly likely to invade important blood vessels during treatment and might cause fatal massive hemorrhage;
11. Patients who have bleeding tendency with abnormal blood coagulation (PT>16s, APTT>43s, TT>21s, Fbg<2g/L); patients treated with anticoagulant or vitamin K antagonists such as warfarin, heparin or its analogues, use a small dose of warfarin (1 mg orally once daily) or a small dose of aspirin (with a daily dose of no more than 100 mg) for prophylactic purposes under the premise of prothrombin time international normalized ratio (INR)≤1.5;
12. Arteriovenous thrombosis events occurred in one year ago, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by venous catheterization due to pre-chemotherapy,but healed) and pulmonary embolism;
13. Patients who have a history of psychotropic drug abuse and were unable to give up or have mental disorders;
14. Patients who have a history of immunodeficiency or other acquired or congenital immunodeficiency disorders or organ transplantation;
15. There were concomitant diseases that seriously endanger the safety of patients or affect the completion of the study according to the judgement of the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2.5 months
  progression-free survival

SECONDARY OUTCOMES:
OS | through study completion, an average of 2 year
  overall survival
ORR | through study completion, an average of 2 year
  objective remission rate
DCR | through study completion, an average of 2 year
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Li, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Result] Dutton SJ, Ferry DR, Blazeby JM, Abbas H, Dahle-Smith A, Mansoor W, Thompson J, Harrison M, Chatterjee A, Falk S, Garcia-Alonso A, Fyfe DW, Hubner RA, Gamble T, Peachey L, Davoudianfar M, Pearson SR, Julier P, Jankowski J, Kerr R, Petty RD. Gefitinib for oesophageal cancer progressing after chemotherapy (COG): a phase 3, multicentre, double-blind, placebo-controlled randomised trial. Lancet Oncol. 2014 Jul;15(8):894-904. doi: 10.1016/S1470-2045(14)70024-5. Epub 2014 Jun 17. PMID 24950987